CLINICAL TRIAL: NCT00746408
Title: Study of the Quality of Self-Diagnosis by Headache Patients Getting Tailored Internet Information
Brief Title: Tailored Internet Information Supply for Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Health & Life Sciences University, Tryol (Other)
Collaborators: Bremen University of Applied Sciences (Other)
Responsible Party: Wilfried Honekamp, Health & Life Sciences University Tyrol, Austria
Other Study IDs: GW Diss 3000490
Record Dates: First submitted 2008-09-02; First posted 2008-09-04 (Estimated); Last update posted 2009-06-16 (Estimated); Status verified 2009-06

CONDITIONS: Headache
Keywords: Internet; Information supply; Tailoring; Patient empowerment; Headaches; Consumer Health Information; Information Services; Information Storage and Retrieval; Information Systems
MeSH Terms: conditions — Headache; Patient Participation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (4):
- Main 1: Insurants of the health insurance company BARMER using the prototype to receive expert system guided tailored internet information about the type of headache they suffer from.
  Interventions: Other: Expert system guided tailored information
- Main 2: Insurants of the health insurance company BARMER using search engines and portals to gather internet information about the type of headache they suffer from.
- Online 1: Internet users using the prototype to receive expert system guided tailored internet information about the type of headache they suffer from.
  Interventions: Other: Expert system guided tailored information
- Online 2: Internet users using search engines and portals to gather internet information about the type of headache they suffer from.

INTERVENTIONS:
Other: Expert system guided tailored information — The prototype is realised by a web-based information system. The HTML web-interface guides the user through the search process by querying the information demand. This is done by an integrated expert system. The expert system uses a rule based inference to determine an internal diagnosis. Based on this internal diagnosis the system searches quality labeled websites and presents relevant information to the user.
  Groups: Main 1; Online 1

SUMMARY:
Medical expert systems in combination with portal searching meta-search engines are exploited to provide reliable patient-tailored information. A prototype of a web-based information system has been developed and is to be evaluated. Its aim is to answer the decisive question whether expert system guided internet meta-search provides a better information supply for patients seeking health information online then this is possible by using ordinary search engines or health portals. The research does neither investigate the influence of ethical nor legal aspects of internet health information supply.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 75
* Suffers at least occasionally from headaches
* Has internet access
* Has not obtained a medical diagnosis (concerning this headache) by a physician, yet

Exclusion Criteria:

* Age under 18
* Age over 75
* Does never suffer from headaches
* Has no internet access
* Has already gotten a medical diagnosis for her/his headaches

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All German speaking adults in the German-speaking part of Europe who suffer at least occasionally from headaches and have not been examined (concerning these headaches) by a physician yet.
  * The population of the main study is narrowed down to a heterogeneous group of insurants of a health insurance company.
  * The population of the online study is self-selecting.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2009-01; Primary Completion 2009-09 (Estimated); Study Completion 2009-09 (Estimated)

PRIMARY OUTCOMES:
Conformity of self-diagnosis and medical diagnosis | After medical diagnoses has been received

CONTACTS AND LOCATIONS:
Overall Officials: Wilfried Honekamp, MSc & Dipl.-Inform., Principal Investigator — Health & Life Sciences University Tyrol, Austria; Herwig Ostermann, Dr., Study Director — Health & Life Sciences University Tyrol, Austria; Roland Staudinger, Prof., Study Chair — Health & Life Sciences University Tyrol, Austria
Locations (1):
- Health & Life Sciences University (UMIT), Hall in Tyrol, Tyrol, Austria

REFERENCES:
- [Background] Eysenbach G, Powell J, Kuss O, Sa ER. Empirical studies assessing the quality of health information for consumers on the world wide web: a systematic review. JAMA. 2002 May 22-29;287(20):2691-700. doi: 10.1001/jama.287.20.2691. PMID 12020305
- [Background] Andrew ME, Penzien DB, Rains JC, Knowlton GE, McAnulty RD. Development of a computer application for headache diagnosis: the Headache Diagnostic System. Int J Biomed Comput. 1992 Jul;31(1):17-24. doi: 10.1016/0020-7101(92)90050-3. PMID 1644498
- [Background] Baur C, Deering MJ. Proposed frameworks to improve the quality of health web sites: review. MedGenMed. 2000 Sep 26;2(3):E35. No abstract available. PMID 11104481
- [Background] Bessell TL, McDonald S, Silagy CA, Anderson JN, Hiller JE, Sansom LN. Do Internet interventions for consumers cause more harm than good? A systematic review. Health Expect. 2002 Mar;5(1):28-37. doi: 10.1046/j.1369-6513.2002.00156.x. PMID 11906539
- [Background] Bindels R, Winkens RA, van Wersch JW, Pop P, Hasman A. Comparing assessment of appropriateness of diagnostic tests between a human expert and an automated reminder system. Stud Health Technol Inform. 2000;77:239-43. PMID 11187550
- [Background] Birru MS, Monaco VM, Charles L, Drew H, Njie V, Bierria T, Detlefsen E, Steinman RA. Internet usage by low-literacy adults seeking health information: an observational analysis. J Med Internet Res. 2004 Sep 3;6(3):e25. doi: 10.2196/jmir.6.3.e25. PMID 15471751
- [Background] Buchanan BG, Moore JD, Forsythe DE, Carenini G, Ohlsson S, Banks G. An intelligent interactive system for delivering individualized information to patients. Artif Intell Med. 1995 Apr;7(2):117-54. doi: 10.1016/0933-3657(94)00029-r. PMID 7647838
- [Background] Bull FC, Kreuter MW, Scharff DP. Effects of tailored, personalized and general health messages on physical activity. Patient Educ Couns. 1999 Feb;36(2):181-92. doi: 10.1016/s0738-3991(98)00134-7. PMID 10223022
- [Background] Eysenbach G, Kohler C, Yihune G, Lampe K, Cross P, Brickley D. A metadata vocabulary for self- and third-party labeling of health web-sites: Health Information Disclosure, Description and Evaluation Language (HIDDEL). Proc AMIA Symp. 2001:169-73. PMID 11825174
- [Background] Gagliardi A, Jadad AR. Examination of instruments used to rate quality of health information on the internet: chronicle of a voyage with an unclear destination. BMJ. 2002 Mar 9;324(7337):569-73. doi: 10.1136/bmj.324.7337.569. PMID 11884320
- [Background] Jadad AR, Gagliardi A. Rating health information on the Internet: navigating to knowledge or to Babel? JAMA. 1998 Feb 25;279(8):611-4. doi: 10.1001/jama.279.8.611. PMID 9486757
- [Background] Kopec D, Shagas G, Selman J, Reinharth D, Tamang S. Development of an expert system for differentiating tension type headaches from migraines. Stud Health Technol Inform. 2004;103:81-92. PMID 15747909
- [Background] Norman CD, Skinner HA. eHealth Literacy: Essential Skills for Consumer Health in a Networked World. J Med Internet Res. 2006 Jun 16;8(2):e9. doi: 10.2196/jmir.8.2.e9. PMID 16867972
- [Background] Olesen J. The International Classification of Headache Disorders. Headache. 2008 May;48(5):691-3. doi: 10.1111/j.1526-4610.2008.01121.x. PMID 18471112
- [Background] Olesen J. International Classification of Headache Disorders, Second Edition (ICHD-2): current status and future revisions. Cephalalgia. 2006 Dec;26(12):1409-10. doi: 10.1111/j.1468-2982.2006.01214.x. No abstract available. PMID 17116090
- [Background] De Simone R, Coppola G, Ranieri A, Bussone G, Cortelli P, D'Amico D, d'Onofrio F, Manzoni GC, Marano E, Perini F, Torelli P, Beneduce L, Ciccarelli G, Mea E, Penza P, Ripa P, Sancisi E, Bonavita V. Validation of AIDA Cefalee, a computer-assisted diagnosis database for the management of headache patients. Neurol Sci. 2007 May;28 Suppl 2:S213-6. doi: 10.1007/s10072-007-0779-z. PMID 17508173
- [Background] Walji M, Sagaram S, Sagaram D, Meric-Bernstam F, Johnson C, Mirza NQ, Bernstam EV. Efficacy of quality criteria to identify potentially harmful information: a cross-sectional survey of complementary and alternative medicine web sites. J Med Internet Res. 2004 Jun 29;6(2):e21. doi: 10.2196/jmir.6.2.e21. PMID 15249270
- [Background] Wilkins ST, Navarro FH. Has the Web really empowered health care consumers? The truth is customers may not have changed as much as we think. Mark Health Serv. 2001 Fall;21(3):5-9. PMID 11525141
- [Background] Winker MA, Flanagin A, Chi-Lum B, White J, Andrews K, Kennett RL, DeAngelis CD, Musacchio RA. Guidelines for medical and health information sites on the internet: principles governing AMA web sites. American Medical Association. JAMA. 2000 Mar 22-29;283(12):1600-6. doi: 10.1001/jama.283.12.1600. PMID 10735398
- [Background] Woolf SH, Krist AH, Johnson RE, Wilson DB, Rothemich SF, Norman GJ, Devers KJ. A practice-sponsored Web site to help patients pursue healthy behaviors: an ACORN study. Ann Fam Med. 2006 Mar-Apr;4(2):148-52. doi: 10.1370/afm.522. PMID 16569718
- See also: The study website — http://www.kopfschmerzlotse.de
- See also: University of Applied Sciences Bremen, Germany — http://www.hs-bremen.de